CLINICAL TRIAL: NCT01188642
Title: Effects of Physical Training and Nutrition Education on Adipocytokines in Severely Obese Teenagers
Acronym: OBAPA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: P. Flammarion, Centre Hospitalier Universitaire de Besançon
Other Study IDs: P/2007/64; 2007-A01319-44 (Other: French Health Products Savety Agency)
Record Dates: First submitted 2010-08-17; First posted 2010-08-25 (Estimated); Last update posted 2010-08-25 (Estimated); Status verified 2010-08

CONDITIONS: Healthy; Obesity
Keywords: childhood obesity; adipocytokines; physical exercise; nutrition education
MeSH Terms: conditions — Obesity; Pediatric Obesity; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: obesity lifestyle intervention — physical activity 5 times per week + nutrition education

SUMMARY:
Obesity is now becoming significantly prevalent of an environment characterized by easily available calorics foods combined with sedentary lifestyles. Moreover, it has been demonstrated that obesity is associated with metabolic complications such as disturbed adipocytokines, hormones secreted by adipose tissue. Given these observations, the purpose of this study is to assess the effects of a lifestyle intervention focused on various physical activities and nutrition education on adipocytokines hormones, in severely obese teenagers.

ELIGIBILITY:
Inclusion Criteria:

* to be aged from 12 to 17
* to have a body mass index > 97 percentile for age and gender

Exclusion criteria:

* systemic disease
* endocrine disorder
* syndromic obesity
* subjects receiving medication with a history of recent intercurrent illness

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: obese teenagers
Sampling Method: Non-Probability Sample
Enrollment: 32
Dates: Start 2009-03; Primary Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Adipocytokines (leptin, adiponectin, ghrelin, PAI-1, resistin), based on subject's arterialized capillary blood samples. | during a lifestyle intervention of 9 months

SECONDARY OUTCOMES:
Body weight, body mass index, waist and hip circumference | during a lifestyle intervention of 9 months
Body composition, calculated by a multifrequency bioelectric impedance | during a lifestyle intervention of 9 months
Glycemia and lipids profile, based on subject's arterialized capillary blood samples analysis. | during a lifestyle intervention of 9 months
Insulin resistance, calculated according to the formula of homeostasis model assessment | during a lifestyle intervention of 9 months
Systolic and diastolic blood pressure, measured in millimeters of mercury at the level of the left brachial artery, using an automatic blood pressure monitor. | during a lifestyle intervention of 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Nhu Uyen Nguyen, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Besançon
Locations (1):
- Centre Hospitalier Universitaire, Besançon, France

REFERENCES:
- [Derived] Gueugnon C, Mougin F, Simon-Rigaud ML, Regnard J, Negre V, Dumoulin G. Effects of an in-patient treatment program based on regular exercise and a balanced diet on high molecular weight adiponectin, resistin levels, and insulin resistance in adolescents with severe obesity. Appl Physiol Nutr Metab. 2012 Aug;37(4):672-9. doi: 10.1139/h2012-045. Epub 2012 May 11. PMID 22574715
- [Derived] Gueugnon C, Mougin F, Nguyen NU, Bouhaddi M, Nicolet-Guenat M, Dumoulin G. Ghrelin and PYY levels in adolescents with severe obesity: effects of weight loss induced by long-term exercise training and modified food habits. Eur J Appl Physiol. 2012 May;112(5):1797-805. doi: 10.1007/s00421-011-2154-2. Epub 2011 Sep 11. PMID 21909986